CLINICAL TRIAL: NCT01790828
Title: Post Marketing Surveillance To Observe Safety And Efficacy Of Xyntha 'Registered' In Subjects With Hemophilia A
Brief Title: Post Marketing Surveillance To Observe Safety And Efficacy Of Xyntha® In Subjects With Hemophilia A
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1831078
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; recombinant factor VIII SQ

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Xyntha group: Xyntha will be administered according to physician's discretion.
  Interventions: Drug: Xyntha : coagulation factor IIIV (recombinant)

INTERVENTIONS:
Drug: Xyntha : coagulation factor IIIV (recombinant) — Xyntha will be administered according to physician's discretion.
  Other Names: Xyntha, MOROCTOCOG ALFA

SUMMARY:
This study is to describe the safety and efficacy of Xyntha® during the usual care setting.

DETAILED DESCRIPTION:
non probability sample

ELIGIBILITY:
Inclusion Criteria:

* Patients or legally authorized representatives of pediatric patients agree to provide written informed consent form (data privacy statement).
* Pediatric and adult patients who have been treated with Xyntha for Hemophilia A from first approved date by KFDA, or who are planned to be newly prescribed Xyntha.

Exclusion Criteria:

* Patients with a known history of hypersensitivity to original or reformulated Xyntha or any component of the product.
* Patients with a known history of hypersensitivity to hamster protein.
* Patients participating in an interventional trial of any investigational drug or device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- South Korea (4):
  - Yonsei Rehabilitation Clinic, Guro-gu, Seoul
  - Kim Hugh Chul Internal Medicine Clinic, Songpa-gu, Seoul
  - Pusan National University Hospital, Busan
  - Kyung Hee University Hospital at Gangdong, Seoul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1831078&StudyName=Post%20Marketing%20Surveillance%20To%20Observe%20Safety%20And%20Efficacy%20Of%20Xyntha%AE%20In%20Subjects%20With%20Hemophilia%20A

RESULTS

PARTICIPANT FLOW:
Groups:
- Xyntha: Non-interventional, observational study of participants who were prescribed and received at least 1 dose of Xyntha 250, 500, 1000, or 2000 IU.
Period: Overall Study
Arm/Group | Xyntha
Started | 42
Completed | 8
Not Completed | 34
Not completed — Other | 34

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Xyntha
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (14.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants by Family History of Factor VIII Inhibitor
Time Frame: 4 years
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Xyntha
Number analyzed (Participants) | 42
percentage of participants
  Yes | 0
  No | 100.0

2. Secondary Outcome: Number of Xyntha Infusions Used to Treat Each New Bleed for On-Demand Therapy (All Participants)
Time Frame: 4 years
Population: All enrolled participants; only participants who received on-demand therapy were included in the analysis.
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | Xyntha
Number analyzed (Participants) | 5
infusions | 1.40 (0.55)

3. Secondary Outcome: Number of Xyntha Infusions Used to Treat Each New Bleed for On-Demand Therapy in Participants Less Than (<)18 Years of Age
Time Frame: 4 years
Population: All enrolled participants; only participants aged <18 years who received on-demand therapy were included in the analysis.
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | Xyntha
Number analyzed (Participants) | 1
infusions | 1.00 (0)

4. Secondary Outcome: Number of Xyntha Infusions Used to Treat Each New Bleed for On-Demand Therapy in Participants Greater Than or Equal to (≥) 18 Years of Age
Time Frame: 4 years
Population: All enrolled participants; participants aged ≥18 years who received on-demand therapy were included in the analysis.
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | Xyntha
Number analyzed (Participants) | 4
infusions | 1.50 (0.58)

5. Secondary Outcome: Number of Responses by Type of Response for All Xyntha Infusions for Treatment of a Bleed for On-Demand Therapy (All Participants)
Description: Response categories were excellent, good, moderate, or no response.
Time Frame: 4 years
Population: All enrolled participants; only participants who received on-demand therapy were included in the analysis.
Measure: Number; unit: Number of responses
Units Other Than Participants: infusions
Arm/Group | Xyntha
Number analyzed (Participants) | 5
Number analyzed (infusions) | 7
Number of responses
  Excellent | 5
  Good | 2
  Moderate | 0
  No response | 0

6. Secondary Outcome: Number of Responses by Type of Response for All Xyntha Infusions for Treatment of a Bleed for On-Demand Therapy in Participants <18 Years of Age
Description: Response categories were excellent, good, moderate, or no response.
Time Frame: 4 years
Population: All enrolled participants; only participants <18 years who received on-demand therapy were included in the analysis.
Measure: Number; unit: number of responses
Units Other Than Participants: infusions
Arm/Group | Xyntha
Number analyzed (Participants) | 1
Number analyzed (infusions) | 1
number of responses
  Excellent | 1
  Good | 0
  Moderate | 0
  No response | 0

7. Secondary Outcome: Number of Responses by Type of Response for All Xyntha Infusions for Treatment of a Bleed for On-Demand Therapy in Participants ≥18 Years of Age
Description: Response categories were excellent, good, moderate, and no response.
Time Frame: 4 years
Population: All enrolled participants; only participants ≥18 years who receive don-demand therapy were included in the analysis.
Measure: Number; unit: number of responses
Units Other Than Participants: infusions
Arm/Group | Xyntha
Number analyzed (Participants) | 4
Number analyzed (infusions) | 6
number of responses
  Excellent | 4
  Good | 2
  Moderate | 0
  No response | 0

8. Secondary Outcome: Number of Participants With Less-Than-Expected Therapeutic Effect (LETE) for On-Demand Therapy
Description: Less than expected therapeutic effect was defined as a 'no response' rating after each of two successive infusions less than or equl to (≤) 24 hours of on-demand therapy.
Time Frame: 4 years
Population: Data were not analyzed as no participants experienced rating of 'no response'.
Arm/Group | Xyntha
Number analyzed (Participants) | 0

9. Secondary Outcome: Average Infusion Dose Per Bleeding for On-Demand Therapy (All Participants)
Time Frame: 4 years
Population: All enrolled participants; only participants who received on-demand therapy were included in the analysis.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Xyntha
Number analyzed (Participants) | 5
IU | 1997.00 (892.77)

10. Secondary Outcome: Average Infusion Dose Per Bleeding for On-Demand Therapy in Participants <18 Years of Age
Time Frame: 4 years
Population: All enrolled participants; only participants <18 years who received on-demand therapy were included in the analysis.
Measure: Median (Full Range); unit: IU
Arm/Group | Xyntha
Number analyzed (Participants) | 1
IU | 725.00 (892.77) [725.00 to 725.00]

11. Secondary Outcome: Average Infusion Dose Per Bleeding for On-Demand Therapy in Participants ≥18 Years of Age
Time Frame: 4 years
Population: All enrolled participants; only participants ≥18 years who received on-demand therapy were included in the analysis.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Xyntha
Number analyzed (Participants) | 4
IU | 2315.00 (623.00)

12. Secondary Outcome: Percentage of Participants Experiencing Hemorrhages During Prophylaxis
Time Frame: 4 years
Population: All enrolled participants; n (number) equals (=) number of participants with nonmissing values
Measure: Number; unit: percentage of participants
Arm/Group | Xyntha
Number analyzed (Participants) | 41
percentage of participants
  All participants (n=41) | 0
  Participants <18 years (n=4) | 0
  Participants ≥18 years (n=37) | 0

13. Secondary Outcome: Annualized Bleeding Rates During Prophylaxis
Description: Annualized bleeding rate defined as total number of breakthrough bleeds within 48 hours (for prophylaxis purpose) divided by (/) [(total period of date of bleeding)/365.25)]
Time Frame: 4 years
Population: Data were not analyzed as information on breakthrough bleeds within 48 hours was not collected.
Arm/Group | Xyntha
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With LETE Bleeds Within 48 Hours of a Preventive/Prophylaxis Dose of Xyntha
Description: Less than expected therapeutic effect for prophylaxis therapy defined as breakthrough (spontaneous/non-traumatic) bleed wtihin 48 hours of prophylaxis infusion.
Time Frame: 4 years
Population: Data were not analyzed as information on breakthrough bleeds within 48 hours was not collected.
Arm/Group | Xyntha
Number analyzed (Participants) | 0

15. Secondary Outcome: Average Infusion Dose During Prophylaxis (All Participants)
Time Frame: 4 years
Population: All enrolled participants; only participants with nonmissing data were included in the analysis.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Xyntha
Number analyzed (Participants) | 41
IU | 1926.70 (532.90)

16. Secondary Outcome: Average Infusion Dose During Prophylaxis in Participants <18 Years of Age
Time Frame: 4 years
Population: All enrolled participants; only participants <18 years were included in the analysis.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Xyntha
Number analyzed (Participants) | 4
IU | 1243.75 (894.51) [725.00 to 725.00]

17. Secondary Outcome: Average Infusion Dose During Prophylaxis in Participants ≥18 Years of Age
Time Frame: 4 years
Population: All enrolled participants; only participants ≥18 years with nonmissing data were included in the analysis.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Xyntha
Number analyzed (Participants) | 37
IU | 2000.16 (437.59)

18. Secondary Outcome: Total Factor Consumption for On-Demand Therapy and During Prophylaxis (All Participants)
Time Frame: 4 years
Population: All enrolled participants; participants were excluded from the analysis if total number of infusions for prophylaxis was unknown.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Xyntha
Number analyzed (Participants) | 18
IU | 66371.00 (60985.45)

19. Secondary Outcome: Total Factor Consumption for On-Demand Therapy and During Prophylaxis in Participants <18 Years of Age
Time Frame: 4 years
Population: All enrolled participants; only participants <18 years were included in the analysis and participants were excluded from the analysis if total number of infusions for prophylaxis was unknown.
Measure: Median (Full Range); unit: IU
Arm/Group | Xyntha
Number analyzed (Participants) | 1
IU | 2900.00 (894.51) [2900.00 to 2900.00]

20. Secondary Outcome: Total Factor Consumption for On-Demand Therapy and During Prophylaxis in Participants ≥18 Years of Age
Time Frame: 4 years
Population: All enrolled participants; only participants ≥18 years were included in the analysis; participants were excluded from the analysis if total number of infusions for prophylaxis was unknown.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Xyntha
Number analyzed (Participants) | 17
IU | 70104.59 (60704.87)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 6 months after the first administration of Xyntha.
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another subject, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Xyntha
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 10/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xyntha (N=42)
Headache (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis fungal (Skin and subcutaneous tissue disorders) | 1
Renal calculus (Renal and urinary disorders) | 1
Xerophthalmia (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No